CLINICAL TRIAL: NCT07282990
Title: Evolution of Endometriosis Lesions and Quality of Life of Patients
Brief Title: Evolution of Endometriosis Lesions Followed by Ultrasound and Quality of Life of Patients: Factors That Influence Disease Progression in a Prospective Cohort
Status: Not yet recruiting | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, Aina Delgado Morell, Co-Investigator, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Other Study IDs: IIBSP-ECE-2024-127
Record Dates: First submitted 2025-12-01; First posted 2025-12-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Endometriosis
Keywords: Endometriosis; Ultrasound; QoL; Progression; Ovarian reserve
MeSH Terms: conditions — Endometriosis; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood (serum and plasma), urine. Endometriosic tissue if surgical exeresis is performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women diagnosed with endometriosis, referred for treatment and/or follow-up to Reference Unit: The study population consists of adult women (18 years or older) with a confirmed diagnosis of endometriosis based on transvaginal ultrasound showing clearly visible and measurable lesions (endometriomas or deep endometriotic lesions suitable for evaluation and follow-up), who are referred for a first consultation at the Endometriosis Reference Unit in Hospital Sant Pau.
  Patients must not have an expected indication for surgical intervention within the next two years, ensuring stable monitoring of disease progression and treatment effects.

SUMMARY:
The goal of this prospective cohort study is to determine the factors that influence the progression of endometriosis and the quality of life of patients.

The main questions it aims to answer are:

1. Is endometriosis a progressive disease?
2. Is the progression of lesions visualized by ultrasound dependent on the medical treatment received?
3. Does the clinical progression of patients correlate with the progression of lesions visualized on transvaginal ultrasound?
4. Is ultrasound follow-up necessary for patients?
5. Could clinical follow-up alone be safe for selected patients?

Researchers will follow up a prospective cohort of 100 patients diagnosed with deep infiltrating endometriosis (DIE) +/- endometriomas during 2 years, collecting data regarding their ultrasound exam and their symptoms and quality of life at stablished controls at recruitment, 6 months, 12 months and 24 months.

DETAILED DESCRIPTION:
This prospective observational cohort study aims to characterize the clinical and ultrasonographic progression of endometriosis and to identify the factors associated with disease evolution, ovarian reserve, symptom burden, and patient-reported quality of life. The protocol is designed to integrate longitudinal clinical assessments, structured transvaginal ultrasound evaluations, hormonal profiling, and digital monitoring through the validated mobile application "Endometric".

The study will follow a cohort of adult women with confirmed endometriosis for two years, using standardized evaluation intervals (baseline, 6 months, 1 year, and 2 years) to capture meaningful changes in lesion morphology, symptoms, and functional outcomes.

Ultrasound assessments will be performed according to the IDEA consensus (Guerriero S, et al. Systematic approach to sonographic evaluation of the pelvis in women with suspected endometriosis, including terms, definitions and measurements: a consensus opinion from the International Deep Endometriosis Analysis (IDEA) group. Ultrasound Obstet Gynecol. 2016 Sep;48(3):318-32. doi: 10.1002/uog.15955) and lesions will be classified using the Enzian system (Keckstein J, et al. The #Enzian classification: A comprehensive non-invasive and surgical description system for endometriosis. Acta Obstet Gynecol Scand. 2021 Jul;100(7):1165-75. doi: 10.1111/aogs.14099), enabling precise measurement of endometriomas, deep infiltrating lesions, associated adhesions, and adnexal involvement.

Ovarian reserve will be estimated using antral follicle count and antimüllerian hormone (AMH) levels, analyzed in a single specialized laboratory to minimize inter-assay variability. Clinical progression will be assessed through standardized symptom scales and the Endometriosis Health Profile Questionnaire (EHP-30). Participants will be managed with expectant, medical, or combined approaches according to routine clinical practice; treatments will not be randomized, but exposure will be precisely documented to evaluate its relationship with disease evolution.

The study functions as a patient registry with predefined longitudinal data collection and structured quality-assurance procedures. Data will be stored in a dedicated Clinapsis database with controlled access and pseudonymization through unique patient codes. A detailed data dictionary will define each variable, its source, coding strategy (including standardized terminology for medications and symptoms), and reference ranges for biological parameters. Automated data-entry checks will detect inconsistencies, missing fields, and out-of-range values at the point of entry. Additional validation procedures will include periodic cross-checks between electronic case-report forms and source data (ultrasound measurements, laboratory results, medical records). Source data verification will be conducted by authorized investigators to ensure accuracy and completeness.

Standard Operating Procedures (SOPs) will govern all registry operations: patient identification and recruitment; informed-consent procedures; clinical and ultrasound assessments; biological-sample handling; data entry, monitoring, and auditing; management of adverse events; and change-control processes for any protocol modifications. The biobank procedures-collection and storage of serum, plasma, urine, and endometriotic tissue-adhere to institutional and regulatory standards, allowing future biomarker research on inflammation, interleukins, and miRNAs.

The planned sample size of 100 patients represents a pragmatic estimate based on available annual referrals and expected retention; although formal power calculations are limited by absent prior data, this cohort is considered sufficient to detect clinically meaningful trends and associations.

Missing data will be addressed through predefined rules distinguishing "missing," "not applicable," and "uninterpretable" entries, with sensitivity analyses planned to assess potential bias.

The statistical analysis plan includes descriptive analysis of all variables according to their scale, repeated-measures ANOVA to evaluate temporal changes across the four scheduled visits, and ANCOVA models to explore the impact of covariates such as age, baseline symptom severity, and treatment type. Comparisons between treatment groups will adjust for confounding when possible, acknowledging that therapeutic choice is not randomized. A significance threshold of 0.05 (two-sided) will be used. Data will be analyzed using IBM SPSS v29 or later.

Monitoring and audit procedures ensure compliance with regulatory and ethical standards. Investigators will maintain study documents for at least five years, and authorized monitors, auditors, ethical committees, or health authorities may access anonymized source documentation for verification.

The project is supported by the Fundació La Marató de TV· (Reg 55/173, project 20241910), which ensures adequate resources for data management, sample processing, and technological support for the clinical-monitoring application.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a confirmed diagnosis of endometriosis, based on ultrasound criteria. Diagnosis must be confirmed by transvaginal ultrasound with evidence of visible and measurable endometriotic lesions.
2. Patients over 18 years of age. This criterion ensures that participants can provide informed consent and are of reproductive age, when the effects of endometriosis and its treatments are relevant to the study.
3. A transvaginal ultrasound performed prior to enrollment showing endometriotic lesions (either endometriomas or deep lesions) with sufficient dimensions and characteristics for evaluation and follow-up.
4. Patients who do not have an indication for scheduled surgery within the next two years. This ensures that the effects of treatment and the progression of the disease can be evaluated throughout the study follow-up period.
5. Signed informed consent from the patient, indicating that she has understood the purpose of the study, the procedures involved, and the potential risks.

Exclusion Criteria:

1. Patients with an indication for scheduled surgical treatment within the next two years. This includes patients requiring surgery for the removal of endometriotic lesions or to address related complications.
2. Patients who are unwilling to undergo follow-up transvaginal ultrasound at scheduled visits (6 months, 1 year, 2 years). Ultrasound is essential for assessing disease progression and the impact of treatment.
3. Patients who are unwilling to participate in the study after receiving all the information and providing their informed consent. Voluntary participation is crucial for the ethics of the study.
4. Patients with intellectual disabilities or conditions that impair their understanding of the study terms and procedures, which could affect their ability to provide valid informed consent.
5. Patients who are pregnant or breastfeeding at the time of enrollment. These conditions can influence the course of endometriosis and the response to treatment, and could complicate disease monitoring.
6. Patients with serious concurrent illnesses or medical conditions that may interfere with the assessment of endometriosis, its progression, or the impact of treatment (e.g., severe chronic inflammatory diseases or cancer).
7. Patients receiving concurrent treatments not permitted by the study protocol (e.g., experimental treatments for endometriosis or related conditions) that may interfere with the interpretation of the results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who are referred to Hospital de la Santa Creu i Sant Pau (Barcelona) due to a clinical or sonographic suspicion of endometriosis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Ultrasound-assessed progression of endometriosic lesions at recruitment, 6, 12 and 24 months | From enrollment to the end of follow-up at 24 months
  * Ultrasound data used:
    * Number of lesions (endometriomas and DIE lesions).
    * Size (assessed in mm; 3 diameters) and characteristics of endometriomas and DIE lesions (described according to IDEA criteria).
    * Presence or absence of hydronephrosis, adhesions, and hydrosalpinx.
  * Ultrasound classification according to Enzian Clssification.
  Outcome variable: PROGRESSION, STABILITY or REGRESSION.
  This result will be defined as follows:
  * PROGRESSION: Increase of > 5mm in the maximum lesion measurement and/or appearance of new lesions and/or increase of 1 point in any item of the Enzian classification.
  * STABILITY: increase/decrease <5mm in the maximum lesion measurement and same number of identified lesions and no changes in the score of any item of the Enzian classification.
  * REGRESSION: decrease > 5mm in the maximum lesion measurement and/or disappearence of any of the previously described lesions and/or decrease of 1 point in any item of the Enzian classification.
Evolution of clinical presentation at recruitment, 6, 12 and 24 months | From enrollment to the end of follow-up at 24 months
  * Symptoms: numeric pain rating scale (zero is equivalent to no pain and 10 indicates the worst possible pain)
    * Dysmenorrhea
    * Chronic pelvic pain
    * Dyschezia
    * Dyspareunia
    * Dysuria
  * Subjective evolution according to patient impressions: Likert scale ("significant improvement" / "moderate improvement" / "stability" / "mild worsening" / "significant worsening")

SECONDARY OUTCOMES:
Evolution of Ovarian Reserve at recruitment, 6, 12 and 24 months | From enrollment to the end of follow-up at 24 months
  Measures:
  * Anti-Müllerian Hormone (AMH) serum level (at first visit and follow-up).
  * Antral Follicle Count (AFC) assessed by transvaginal ultrasound (at first visit and follow-up).
  Outcome variable: OVARIAN RESERVE LOSS (YES / NO) Decreased ovarian reserve will be considered when AMH presents with a drop of 0.2 ng/mL annually, and/or if AMH if below 1 ng/dL at any time during follow-up, and/or AFC falls >=4 follicles anually.
Evolution of Quality of Life (QoL) at recruitment, 6, 12 and 24 monts | From enrollment to the end of follow-up at 24 months
  - Quality of life measurement using the Endometriosis Health Profile-30 (EHP-30) questionnaire (at first visit and follow-up).
  The EHP-30 consists of a core instrument which includes five scale scores covering:
  * Pain (11 items)
  * Control and powerlessness (6 items)
  * Social support (4 items)
  * Emotional well-being (6 items)
  * Self-image (3 items)
  Each item is answered as a categorical Likert-Scale (Never, Rarely, Sometimes, Often, Always).
  It is a self-reported questionnaire which will be administered on paper support.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying the results will be shared in a deidentified format for research purposes.
  Supporting Documents: Study protocol, statistical analysis plan, and informed consent form will also be available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available beginning 6-12 months after publication of the primary results and will remain accessible for at least 5 years.
Access Criteria: Data will be shared with qualified researchers upon reasonable request sent to study IP.
  Access will require a data-sharing agreement ensuring appropriate use, data protection, and compliance with ethical standards.

REFERENCES:
- [Background] Vannuccini S, Clemenza S, Rossi M, Petraglia F. Hormonal treatments for endometriosis: The endocrine background. Rev Endocr Metab Disord. 2022 Jun;23(3):333-355. doi: 10.1007/s11154-021-09666-w. Epub 2021 Aug 17. PMID 34405378
- [Background] Brown J, Crawford TJ, Datta S, Prentice A. Oral contraceptives for pain associated with endometriosis. Cochrane Database Syst Rev. 2018 May 22;5(5):CD001019. doi: 10.1002/14651858.CD001019.pub3. PMID 29786828
- [Background] Vercellini P, Crosignani P, Somigliana E, Vigano P, Frattaruolo MP, Fedele L. 'Waiting for Godot': a commonsense approach to the medical treatment of endometriosis. Hum Reprod. 2011 Jan;26(1):3-13. doi: 10.1093/humrep/deq302. Epub 2010 Nov 11. PMID 21071490
- [Background] Becker CM, Bokor A, Heikinheimo O, Horne A, Jansen F, Kiesel L, King K, Kvaskoff M, Nap A, Petersen K, Saridogan E, Tomassetti C, van Hanegem N, Vulliemoz N, Vermeulen N; ESHRE Endometriosis Guideline Group. ESHRE guideline: endometriosis. Hum Reprod Open. 2022 Feb 26;2022(2):hoac009. doi: 10.1093/hropen/hoac009. eCollection 2022. PMID 35350465
- [Background] National Guideline Alliance (UK). Endometriosis: diagnosis and management. London: National Institute for Health and Care Excellence (NICE); 2017 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK453273/ PMID 29787038
- [Background] Koninckx PR, Fernandes R, Ussia A, Schindler L, Wattiez A, Al-Suwaidi S, Amro B, Al-Maamari B, Hakim Z, Tahlak M. Pathogenesis Based Diagnosis and Treatment of Endometriosis. Front Endocrinol (Lausanne). 2021 Nov 25;12:745548. doi: 10.3389/fendo.2021.745548. eCollection 2021. PMID 34899597
- [Background] de Ziegler D, Borghese B, Chapron C. Endometriosis and infertility: pathophysiology and management. Lancet. 2010 Aug 28;376(9742):730-8. doi: 10.1016/S0140-6736(10)60490-4. PMID 20801404
- [Background] Perello MF, Martinez-Zamora MA, Torres X, Munros J, Balasch Cortina J, Carmona F. Endometriotic Pain Is Associated with Adenomyosis but Not with the Compartments Affected by Deep Infiltrating Endometriosis. Gynecol Obstet Invest. 2017;82(3):240-246. doi: 10.1159/000447633. Epub 2016 Oct 7. PMID 27710968
- [Background] Chamie LP, Ribeiro DMFR, Tiferes DA, Macedo Neto AC, Serafini PC. Atypical Sites of Deeply Infiltrative Endometriosis: Clinical Characteristics and Imaging Findings. Radiographics. 2018 Jan-Feb;38(1):309-328. doi: 10.1148/rg.2018170093. PMID 29320327
- [Background] Koninckx PR, Ussia A, Adamyan L, Wattiez A, Donnez J. Deep endometriosis: definition, diagnosis, and treatment. Fertil Steril. 2012 Sep;98(3):564-71. doi: 10.1016/j.fertnstert.2012.07.1061. PMID 22938769
- [Background] Koninckx PR, Ussia A, Adamyan L, Tahlak M, Keckstein J, Wattiez A, Martin DC. The epidemiology of endometriosis is poorly known as the pathophysiology and diagnosis are unclear. Best Pract Res Clin Obstet Gynaecol. 2021 Mar;71:14-26. doi: 10.1016/j.bpobgyn.2020.08.005. Epub 2020 Sep 1. PMID 32978068
- [Background] Chapron C, Marcellin L, Borghese B, Santulli P. Rethinking mechanisms, diagnosis and management of endometriosis. Nat Rev Endocrinol. 2019 Nov;15(11):666-682. doi: 10.1038/s41574-019-0245-z. Epub 2019 Sep 5. PMID 31488888
- [Background] De Graaff AA, D'Hooghe TM, Dunselman GA, Dirksen CD, Hummelshoj L; WERF EndoCost Consortium; Simoens S. The significant effect of endometriosis on physical, mental and social wellbeing: results from an international cross-sectional survey. Hum Reprod. 2013 Oct;28(10):2677-85. doi: 10.1093/humrep/det284. Epub 2013 Jul 11. PMID 23847114
- [Background] Keckstein J, Saridogan E, Ulrich UA, Sillem M, Oppelt P, Schweppe KW, Krentel H, Janschek E, Exacoustos C, Malzoni M, Mueller M, Roman H, Condous G, Forman A, Jansen FW, Bokor A, Simedrea V, Hudelist G. The #Enzian classification: A comprehensive non-invasive and surgical description system for endometriosis. Acta Obstet Gynecol Scand. 2021 Jul;100(7):1165-1175. doi: 10.1111/aogs.14099. Epub 2021 Mar 19. PMID 33483970
- [Background] Giudice LC, Kao LC. Endometriosis. Lancet. 2004 Nov 13-19;364(9447):1789-99. doi: 10.1016/S0140-6736(04)17403-5. PMID 15541453